CLINICAL TRIAL: NCT01022333
Title: The Potential for Oral DIM Supplementation to Increase the Production of the BRCA1 Protein in BRCA1 Mutation Carriers
Brief Title: The Potential for Oral Diindolylmethane (DIM) Supplementation to Increase the Production of the BRCA1 Protein in BRCA1 Mutation Carriers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women's College Hospital (Other)
Collaborators: BioResponse (Industry)
Responsible Party: Dr. Steven A. Narod, MD, Familial Breast Cancer Research Unit, Women's College Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2009-015-B
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Breast Cancer
Keywords: BRCA1; breast cancer; 3,3'-di-indolylmethane; dietary intervention; estrogen metabolites; mRNA expression; BRCA1 protein; Estrogen
MeSH Terms: conditions — Breast Neoplasms | interventions — 3,3'-diindolylmethane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DIM group (BRCA1 carriers) (Experimental): This group will have up to 100 women who are carriers of a BRCA1 deleterious mutation. To ensure safety, women in this group will not be able to participate in the study if they are under medications with warfarin, theophylline, or anticonvulsants; or if they are pregnant, breast-feeding or planning to become pregnant within 6 months of the research project. Women in this group will receive 300 mg per day of Rx Balance BioResponse DIM for six weeks. Supplements will be given free of charge. A blood sample (20cc) and a urine sample (20cc) will be collected from these women during two clinic visits; the second visit will be during the six weeks of DIM supplementation (4-6 weeks after the first clinic visit).
  Interventions: Dietary Supplement: Diindolylmethane (DIM)
- No DIM group (BRCA1 carriers) (No Intervention): This group will have up to a 100 women who are carriers of a BRCA1 deleterious mutation. This group will not receive DIM. Women that choose not to take DIM will be in this group. A blood sample (20cc) and a urine sample (20cc) will be collected from these women during two clinic visits; the second visit will be 4-6 weeks after the first clinic visit.
- General Control Group (No Intervention): This group will have up to 100 women who do not carry a BRCA1 mutation but who come from BRCA1 carrier family (a family with at least one individual that has tested positive for a BRCA1 mutation). A control subject is considered negative for a BRCA1 mutation if she has been confirmed by direct DNA sequencing to not be a carrier of this gene. A blood sample (20cc) and a urine sample (20cc) will be collected from these women at a single clinic visit.

INTERVENTIONS:
Dietary Supplement: Diindolylmethane (DIM) — 300 mg per day of DIM for six weeks.
  Other Names: Rx Balance BioResponse DIM
  Arms: DIM group (BRCA1 carriers)

SUMMARY:
Women with a BRCA1 mutation face a lifetime risk of breast cancer of approximately 70% and a lifetime risk of ovarian cancer of approximately 40%. A number of potential anti-cancer nutrients have been proposed, however, it is important that diet supplements be evaluated prior to general recommendation.

The risk of breast and ovarian cancer in carriers of a BRCA1 mutation might be lowered by some nutritional supplements. For example, green tea, broccoli and vitamin D are of potential interest. One dietary supplement that is thought to have potential for BRCA1 carriers is diindolylmethane (DIM), which is an active ingredient in broccoli and other green vegetables. DIM - is found in vegetables like broccoli and is available as a supplement in health food stores. The investigators think that DIM may increase the production of the normal copy of BRCA1 and offset the effect of the mutation.

The purpose of this study is to determine that there is a potential for oral DIM supplementation to result in the increased production of the BRCA1 protein in BRCA1 mutation carriers. The results of the study will also serve as an evaluation of the current use and success of preventive strategies for BRCA1 mutation carriers.

ELIGIBILITY:
Inclusion Criteria:

* Carriers of a mutation in the BRCA1 gene
* Non-carriers of a mutation in the BRCA1 gene who come from a family with a BRCA1 mutation (a family in which at least one individual has tested positive for a BRCA1 mutation)
* Can participate after being free of DIM supplementation for one month

Exclusion Criteria:

* Have a personal history of cancer
* Currently pregnant or breast-feeding

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-07 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Oral DIM supplementation increases BRCA1 mRNA expression and hence BRCA1 protein in women with a BRCA1 mutation | 6 months

SECONDARY OUTCOMES:
Oral DIM supplementation causes favorable estrogen metabolism in women with a BRCA1 mutation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Narod, MD, Principal Investigator — Women's College Research Institute
Locations (1):
- Familial Breast Cancer Research Unit, Women's College Research Institute, Toronto, Ontario, Canada